CLINICAL TRIAL: NCT05857384
Title: A Randomised Four-Period Cross-Over Phase I Study to Assess Bioavailability, Bioequivalence and Tolerability of IHL-42X Compared to the Reference Drugs in Healthy Volunteers
Brief Title: Bioavailability, Bioequivalence and Tolerability of IHL-42X Compared to the Reference Drugs
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Incannex Healthcare Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IHL42XBABE
Record Dates: First submitted 2023-02-27; First posted 2023-05-12 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-11

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Acetazolamide; Dronabinol

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (4):
- Comparator Arm A- Reference Listed Drug/Marinol (Active Comparator): dronabinol 5 mg, two capsules of 2.5 mg administered on an empty stomach once only in the study period
  Interventions: Drug: Dronabinol 2.5 MG
- Comparator Arm B-Reference Listed Drug/Taro Acetazolamide (Active Comparator): 250 mg acetazolamide, one tablet administered on an empty stomach once only in the study period
  Interventions: Drug: Acetazolamide 250 MG
- Investigational Product Arm C-IHL42X Fasted (Experimental): IHL-42X (5 mg dronabinol, 250 mg acetazolamide), one capsule administered on an empty stomach once only in the study period
  Interventions: Drug: IHL42X
- Investigational Product Arm D-IHL42X Fed (Experimental): IHL-42X (5 mg dronabinol, 250 mg acetazolamide), one capsule administered after food once only in the study period
  Interventions: Drug: IHL42X

INTERVENTIONS:
Drug: IHL42X — IHL-42X consists of acetazolamide and dronabinol.
  Other Names: IHL-42X
  Arms: Investigational Product Arm C-IHL42X Fasted; Investigational Product Arm D-IHL42X Fed
Drug: Acetazolamide 250 MG — A solid tablet containing 250 mg acetazolamide
  Other Names: Taro Acetazolamide
  Arms: Comparator Arm B-Reference Listed Drug/Taro Acetazolamide
Drug: Dronabinol 2.5 MG — A soft gelatin capsules containing 2.5mg dronabinol
  Other Names: Marinol
  Arms: Comparator Arm A- Reference Listed Drug/Marinol

SUMMARY:
The goal of this randomised four-period cross-over Phase I study is to assess bioavailability, bioequivalence and tolerability of IHL-42X compared to the reference drugs in healthy volunteers.

Volunteers will be enrolled and randomised to one of four treatment groups. Each group is to receive all four treatments in a twenty eight day cross-over study, with each treatment period running for seven days.

The four treatment groups are described below; A = dronabinol 5 mg, fasted; B = acetazolamide 250 mg, fasted; C = IHL-42X (5 mg dronabinol, 250 mg acetazolamide), fasted; D = IHL-42X (5 mg dronabinol, 250 mg acetazolamide), fed. Each treatment group will enrol at least 29 participants each, for a total of at least 116 participants.

Bioavailability and bioequivalence will assess and compare all four of the seven day treatments.

DETAILED DESCRIPTION:
This is a 4-period crossover bioequivalence and bioavailability clinical trial designed to assess the pharmacokinetics and safety and tolerability of IHL-42X compared to the reference listed drugs Marinol (reference listed drug for dronabinol) and Taro acetazolamide (reference listed drug for acetazolamide). The study will look to enrol at least 116 participants. Participants will be enrolled into one of four treatment groups, each group consisting of approximately 29 participants, which will receive all four treatments in different orders, as defined by period 1, period 2, period 3 and period 4.

The trial will recruit healthy participants if they satisfy all the following criteria:

1. Ages ≥18 to ≤65 at the time of screening
2. BMI ≥18.0 to ≤32.0
3. Physically well, in the opinion of the investigator, with no clinically significant psychiatric, cardiac, hepatic, renal, endocrine, gastrointestinal, bleeding, thyroid, cholesterol, or hypertension disorders
4. If male, willing to use an approved method of contraception from 30 days prior to dosing, throughout the study, and 90 days after last dose.
5. If female of non-childbearing potential, must be postmenopausal with established serum FSH levels >30IU/L (determined during screening or have undergone one of the sterilization procedures, as noted in the protocol, at least 6 months prior to Visit Day 1 If females of childbearing potential, must not be currently pregnant, lactating, or planning to be pregnant and are willing to use an approved method of contraception, as noted in the protocol, from 30 days prior to dosing, throughout the study, and 30 days after last dose. Partner has had a vasectomy at least 6 months prior to first dose Of non-childbearing potential (postmenopausal or surgically sterile by any method for at least 3 months prior to check-in) Abstinence Same sex relationship
6. Voluntarily consent to participate in the study and complete all study required tasks, as instructed by the protocol, including the completion of questionnaires.

Participants will be excluded from participating in the study if there is evidence of any of the following at screening, or prior to dosing at the timepoints in the Schedule of Events:

1. History of cardiac disease or arrythmias
2. History of significant psychiatric illness (defined as hospitalisation or history of pharmacological prescription for psychiatric conditions), suicidal ideation, or suicidal attempts
3. Current use of illicit drugs or as defined by a positive urine drug test at screening or baseline
4. History of alcohol abuse or excessive alcohol intake according to the Australian guidelines (more than 10 standard drinks per week/4 standard drinks per day on average) or alcohol consumption (by self-declaration) defined as > 21 alcohol units per week (where 1 unit = 284 mL of beer, 25 mL of 40% spirit, or a 125 mL glass of wine).
5. Any cannabis use within 30 days of screening
6. Known hypersensitivity and/or intolerance to any cannabis products with previous use
7. Known hypersensitivity and/or intolerance to sesame oil (dronabinol is formulated in sesame oil)
8. Known hypersensitivity and/or intolerance to acetazolamide
9. Has taken any vitamins, herbal remedies, supplements or cannabidiol products within 7 days of each check-in
10. GAD-7 score of ≥15, MDI score ≥31 OR 3 core symptoms and 5 accompanying symptoms, C-SSRS score ≥4 OR reported suicidal behaviour within the past 3 months
11. Any dietary requirements incompatible with study breakfast; must be able to eat high- fat, high-calorie diet (including meat, dairy products) (As described in FDA guidance for BA and BE studies (See Appendix 6 in protocol))
12. Hepatic or renal impairment or disease, as defined as AST/ALT >1.5 x ULN, eGFR <60 at screening and check-in.
13. History of gastrointestinal disorders or previous surgeries which may impact absorption, distribution, metabolism and/or excretion of the IP (such as cholecystitis, cholecystectomy)
14. Female participants who are pregnant, lactating or planning to become pregnant
15. Inability to adhere to the protocol and study restrictions during the study period
16. Participation in another clinical trial of an investigational drug within 30 days or 5 half- lives of the investigational drug (whichever is longer) prior to first study drug administration.
17. Any other reason in the opinion of the investigator

During the 28-day screening period, participants will provide information on their demographics, medical history, height, weight and BMI. A physical exam, vital signs and 12-lead ECG will be conducted. Blood and urine tests will be performed to ensure there are no clinically significant outcomes that would exclude the participants from enrolling in the study, and urine will be tested for pregnancy and for the presence of illicit drugs. Questionnaires to review mental health status of the participants will also be conducted. These will include the General Anxiety Disorder -7 (GAD-7), Major Depression Index (MDI) and the Columbia Suicide Severity Rating Scale (C-SSRS).

Once the participant is deemed eligible to be enrolled in the study, the baseline visit will be performed and the participant will be randomised into one of the four groups and will receive each of the four treatments in the order, as described below:

Participants randomised to Group 1 will receive treatments in the following order:

Group 1 - A, B, C D

Participants randomised to Group 2 will receive treatments in the following order:

Group 2 - B, D, C, A

Participants randomised to Group 3 will receive treatments in the following order:

Group 3 - C, A, D, B

Participants randomised to Group 4 will receive treatments in the following order:

Group 4 - D, C, B, A,

where; Treatment Group A = dronabinol 5 mg, fasted; Treatment Group B = acetazolamide 250 mg, fasted; Treatment Group C = IHL-42X (5 mg dronabinol, 250 mg acetazolamide), fasted; Treatment Group D = IHL-42X (5 mg dronabinol, 250 mg acetazolamide), fed.

The participant will stay in the clinic for each of the treatment periods. Assessments include vital signs, 12-lead ECG, urine and blood sampling and testing will be repeated. Depending on the randomisation group, the participant will receive one dose of the treatment. Blood draws for pharmacokinetics will be conducted and the participant monitored for adverse events.

For treatment groups A, B and C, the participant will fast for 10 hours prior to receiving the dose of either dronabinol, acetazolamide or IHL-42X. For treatment group D, the participant will be required to consume a high fat/high calorie diet 30 minutes prior to receiving the dose of IHL-42X.

Blood samples will be taken for pharmacokinetics analysis throughout the study, at specific timepoints, including on prior to dosing. These samples will be assessed for THC and acetazolamide, as well as the metabolites of THC.

Participants will be discharged from the clinic on day 3 of each period, at least 48 hours post dose, and will return to the clinic after a minimum of 7 days, to allow for washout, from the dose date to begin the next treatment period.

The last dose timepoint assessments at 48 hours post final dose for period 4 will serve as the end of study visit.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers will be enrolled in the study if they satisfy all the following criteria:

  1. Ages ≥18 to ≤65 at the time of screening
  2. BMI ≥18.0 to ≤32.0
  3. Physically well, in the opinion of the investigator, with no clinically significant psychiatric, cardiac, hepatic, renal, endocrine, gastrointestinal, bleeding, thyroid, cholesterol, or hypertension disorders
  4. If male, willing to use an approved method of contraception from 30 days prior to dosing, throughout the study, and 90 days after last dose.

     Options include:

     Surgically sterile (vasectomy at least 6 months prior to dosing) Condom + partner with IUD device (in place 3 months prior to dosing through to 90 days after last dose) Condom + partner with diaphragm for at least 30 days prior to dosing through to 90 days after last dose Condom + partner using hormonal contraception for at least 3 months prior to dosing + condom for at least 30 days prior to dosing through to 90 days after last dose OR Contraception not required Sexual partner is surgically sterile. Partner is of non-childbearing potential Same sex relationship Abstinence
  5. If female of non-childbearing potential, must be postmenopausal with established serum FSH levels >30IU/L (determined during screening or have undergone one of the following sterilization procedures at least 6 months prior to Visit Day 1;

     1. Bilateral tubal ligation
     2. Hysterectomy
     3. Hysterectomy with unilateral or bilateral oophorectomy
     4. Bilateral oophorectomy If females of childbearing potential must not be currently pregnant, lactating, or planning to be pregnant and are willing to use an approved method of contraception from 30 days prior to dosing, throughout the study, and 30 days after last dose.

     Options include:

     Condom + IUD device (in place 3 months prior to dosing + 30 days after last dose) Condom + Diaphragm for at least 30 days prior to dosing + 30 days after last dose Condom + Hormonal contraception for at least 3 months prior to dosing + condom for at least 30 days prior to dosing + 30 days after last dose OR Contraception not required Partner has had a vasectomy at least 6 months prior to first dose Of non-childbearing potential (postmenopausal or surgically sterile by any method for at least 3 months prior to check-in) Abstinence Same sex relationship
  6. Voluntarily consent to participate in the study and complete all study required tasks, as instructed by the protocol, including the completion of questionnaires.

Exclusion Criteria:

* Healthy volunteers will be excluded from the study if there is evidence of any of the following at screening, or prior to dosing at the timepoints in the Schedule of Events.

  1. History of cardiac disease or arrythmias
  2. History of significant psychiatric illness (defined as hospitalisation or history of pharmacological prescription for psychiatric conditions), suicidal ideation, or suicidal attempts
  3. Current use of illicit drugs or as defined by a positive urine drug test at screening or baseline
  4. History of alcohol abuse or excessive alcohol intake according to the Australian guidelines (more than 10 standard drinks per week/4 standard drinks per day on average) or alcohol consumption (by self-declaration) defined as > 21 alcohol units per week (where 1 unit = 284 mL of beer, 25 mL of 40% spirit, or a 125 mL glass of wine).
  5. Any cannabis use within 30 days of screening
  6. Known hypersensitivity and/or intolerance to any cannabis products with previous use
  7. Known hypersensitivity and/or intolerance to sesame oil (dronabinol is formulated in sesame oil)
  8. Known hypersensitivity and/or intolerance to acetazolamide
  9. Has taken any vitamins, herbal remedies, supplements or cannabidiol products within 7 days of each check-in
  10. GAD-7 score of ≥15, MDI score ≥31 OR 3 core symptoms and 5 accompanying symptoms, C-SSRS score ≥4 OR reported suicidal behaviour within the past 3 months
  11. Any dietary requirements incompatible with study breakfast; must be able to eat high-fat, high-calorie diet (including meat, dairy products) (As described in FDA guidance for BA and BE studies (Appendix 6))
  12. Hepatic or renal impairment or disease, as defined as AST/ALT >1.5 x ULN, eGFR <60 at screening and check-in.
  13. History of gastrointestinal disorders or previous surgeries which may impact absorption, distribution, metabolism and/or excretion of the IP (such as cholecystitis, cholecystectomy)
  14. Female participants who are pregnant, lactating or planning to become pregnant
  15. Inability to adhere to the protocol and study restrictions during the study period
  16. Participation in another clinical trial of an investigational drug within 30 days or 5 half-lives of the investigational drug (whichever is longer) prior to first study drug administration.
  17. Any other reason in the opinion of the investigator

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2023-09-08 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Bioavailability of IHL-42X | 28 days
  Assess the proportion of IHL-42X that is taken up and enters the circulation post dose.
Bioequivalence of IHL-42X | 28 days
  Compare the proportion of IHL-42X taken up and enters the circulation to the reference listed drugs for dronabinol and acetazolamide. It will be determined whereby 90% confidence interval for the ratio of averages of measures Cmax and AUC0-inf for IHL-42X and the reference listed drug.
Effect of food on IHL-42X - maximum observed drug concentration | 7 days
  Assess the effect of food on the uptake and absorption of IHL-42X by measuring Cmax (Maximum observed drug concentration)
Effect of food on IHL-42X - time of the maximum drug concentration | 7 days
  Assess the effect of food on the uptake and absorption of IHL-42X by measuring Tmax (time of the maximum drug concentration)
Effect of food on IHL-42X - area under the drug concentration time curve from time zero to time of last measurable concentration | 7 days
  Assess the effect of food on the uptake and absorption of IHL-42X by measuring AUC0-last (Area under the drug concentration-time curve, from time zero to time of last measurable concentration)
Effect of food on IHL-42X - area under the drug concentration time curve from time zero to infinity | 7 days
  Assess the effect of food on the uptake and absorption of IHL-42X by measuring AUC0-inf (Area under the drug concentration-time curve from time zero to infinity)
Effect of food on IHL-42X - area under the drug concentration time curve from time zero to 12 hours | 7 days
  Assess the effect of food on the uptake and absorption of IHL-42X by measuring AUC0-12h (Area under the drug concentration-time curve from time zero to 12 hours)
Effect of food on IHL-42X - area under the drug concentration time curve from time zero to 24 hours | 7 days
  Assess the effect of food on the uptake and absorption of IHL-42X by measuring AUC0-24h (Area under the drug concentration-time curve from time zero to 24 hours)
Effect of food on IHL-42X - the elimination half-life | 7 days
  Assess the effect of food on the uptake and absorption of IHL-42X by measuring t1/2 (the elimination half-life)
Effect of food on IHL-42X - terminal elimination rate constant | 7 days
  Assess the effect of food on the uptake and absorption of IHL-42X by measuring kel (Terminal elimination rate constant)
Effect of food on IHL-42X - apparent total body clearance | 7 days
  Assess the effect of food on the uptake and absorption of IHL-42X by measuring CL/F (Apparent total body clearance)
Effect of food on IHL-42X - apparent volume of distribution | 7 days
  Assess the effect of food on the uptake and absorption of IHL-42X by measuring Vz/F (Apparent volume of distribution)

SECONDARY OUTCOMES:
Safety and tolerability | 28 days
  Assess the number of treatment emergent adverse events (TEAEs) and serious treatment emergent adverse events associated with the dosing of IHL-42X in comparison to the reference listed drugs, dronabinol and acetazolamide.

CONTACTS AND LOCATIONS:
Overall Officials: Emir Redzepagic, MBBS, Principal Investigator — CMAX Clinical Research; Phillip Ryan, MBBS, Principal Investigator — Nucleus Network Pty Ltd.
Locations (4):
- Australia (4):
  - CMAX, Adelaide, South Australia
  - Nucleus Network Pty Ltd, Geelong, Victoria
  - Nucleus Network Pty Ltd [Commercial Road], Melbourne, Victoria
  - Nucleus Network Pty Ltd, Melbourne, Victoria